CLINICAL TRIAL: NCT04753762
Title: Multimodal IMAgery (Echocardiography and Cardiac MRI) Characterization of Cardiac Damage and Severity After COVID-19 Infection
Brief Title: Multimodal IMAgery Characterization of Cardiac Damage and Severity After COVID-19 Infection
Acronym: IMACovid
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Laura FILIPPETTI, Doctor, Central Hospital, Nancy, France
Other Study IDs: 2020PI086
Record Dates: First submitted 2021-01-26; First posted 2021-02-15 (Actual); Last update posted 2023-05-08 (Actual); Status verified 2023-05

CONDITIONS: COVID-19 Virus Disease; Cardiac Complication
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Coronavirus Disease 2019 (COVID-19) is an infection caused by Severe Acute Respiratory Syndrome Coronavirus (SARS-CoV-2), which affects multiple organ system particularly the lung and heart. Indeed, SARS CoV-2 has various cardiac manifestations which are associated with higher mortality and morbidity. Cardiac involvement, based on elevated levels of myocardial enzymes, have been described in 20 to 30% of COVID-19 infection. However, the physiopathological mechanisms of myocardial injury remains unclear. Main hypothesis include inflammation and cytokine storm, hypercoagulability and vascular thrombosis, inflammation or stress leading to coronary plaque rupture (type I myocardial infarction), supply-demand mismatch and hypoxemia resulting in myocardial damage (type II myocardial infarction) ...

Two patterns can be identified : ischemic or non-ischemic pattern including myocarditis, stress induced cardiomyopathy, thrombo-embolic disease. However, the consequences of myocardial damage after confirmed COVID-19 infection are unknown at medium to long term prognosis.

Data are needed to identify myocardial damage and to guide effective therapies and follow-up (use of ACE inhibitor, beta-blockers, steroids...? ) In this study, the investigators proposed to collect multimodal cardiac imaging including MRI (Magnetic Resonance Imaging) and TTE (Transthoracic echocardiogram) in order to identify and characterize cardiac injury as ischemic or non-ischemic pattern, to better assess risk stratification and to guide effective therapies if necessary.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac involvement confirmed : increase troponin level > 50pg/ml or left ventricular dysfunction assessed by echocardiography during hospitalization for confirmed COVID-19 infection
* Absence of severe renal failure (CKD EPI > 30ml/min/1.73m²)
* Cardic imaging (MRI and TTE) performed during 4 months from COVID-19 infection

Exclusion Criteria:

* Cardiovascular history (ischemic or valvular disease, dilated cardiomyopathy, cardiac surgery...)
* Vulnerable patient (pregnancy, adult under legal protection)

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients increase troponin level > 50ng/ml or left ventricular dysfunction assessed by echocardiography during hospitalization for confirmed COVID-19 infection
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
To Characterize cardiac involvement by cardiac TTE imaging during 4 months after confirmed COVID-19 infection | 1 to 4 months after COVID 19 infection
  Cardiac TTE imaging is performed during 4 months after COVID-19 infection in patients with suspected cardiac involvement (increase troponin level>50ng/ml or left ventricular dysfunction during hospitalisation for COVID-19 infection) in order to determine tissular characterization, in particular the presence of ischemic or non-ischemic pattern.
To Characterize cardiac involvement by cardiac MRI during 4 months after confirmed COVID-19 infection | 1 to 4 months after COVID 19 infection
  Cardiac MRI is performed during 4 months after COVID-19 infection in patients with suspected cardiac involvement (increase troponin level>50ng/ml or left ventricular dysfunction during hospitalisation for COVID-19 infection) in order to determine tissular characterization, in particular the presence of ischemic or non-ischemic pattern.

SECONDARY OUTCOMES:
To characterize cardiac evolution at 12 +/-2 months from COVID-19 infection | 12 +/- 2 months
  Cardiac imaging are performed 12 +/-2 months after COVID-19 infection
To evaluate Cardiac events at 12 +/-2 months from COVID-19 infection | 12+/-2 months
  Follow-up at 12+/-2 months from COVID-19 infection :
  - medical consultation to collect cardiac events (heart failure, arrythmias, chest pain).
To evaluate all cause deaths at 12 +/-2 months from COVID-19 infection | 12+/-2 months
  Follow-up at 12+/-2 months from COVID-19 infection :
  - status (dead or alive)

CONTACTS AND LOCATIONS:
Overall Officials: Laura FILIPPETTI, MD, Principal Investigator — CHRU NANCY
Locations (1):
- Laura FILIPPETTI, Vandœuvre-lès-Nancy, France

REFERENCES:
- [Result] Wang D, Hu B, Hu C, Zhu F, Liu X, Zhang J, Wang B, Xiang H, Cheng Z, Xiong Y, Zhao Y, Li Y, Wang X, Peng Z. Clinical Characteristics of 138 Hospitalized Patients With 2019 Novel Coronavirus-Infected Pneumonia in Wuhan, China. JAMA. 2020 Mar 17;323(11):1061-1069. doi: 10.1001/jama.2020.1585. PMID 32031570
- [Result] Bavishi C, Bonow RO, Trivedi V, Abbott JD, Messerli FH, Bhatt DL. Special Article - Acute myocardial injury in patients hospitalized with COVID-19 infection: A review. Prog Cardiovasc Dis. 2020 Sep-Oct;63(5):682-689. doi: 10.1016/j.pcad.2020.05.013. Epub 2020 Jun 6. PMID 32512122
- [Result] Driggin E, Madhavan MV, Bikdeli B, Chuich T, Laracy J, Biondi-Zoccai G, Brown TS, Der Nigoghossian C, Zidar DA, Haythe J, Brodie D, Beckman JA, Kirtane AJ, Stone GW, Krumholz HM, Parikh SA. Cardiovascular Considerations for Patients, Health Care Workers, and Health Systems During the COVID-19 Pandemic. J Am Coll Cardiol. 2020 May 12;75(18):2352-2371. doi: 10.1016/j.jacc.2020.03.031. Epub 2020 Mar 19. PMID 32201335
- [Result] Inciardi RM, Lupi L, Zaccone G, Italia L, Raffo M, Tomasoni D, Cani DS, Cerini M, Farina D, Gavazzi E, Maroldi R, Adamo M, Ammirati E, Sinagra G, Lombardi CM, Metra M. Cardiac Involvement in a Patient With Coronavirus Disease 2019 (COVID-19). JAMA Cardiol. 2020 Jul 1;5(7):819-824. doi: 10.1001/jamacardio.2020.1096. PMID 32219357
- [Result] Babapoor-Farrokhran S, Gill D, Walker J, Rasekhi RT, Bozorgnia B, Amanullah A. Myocardial injury and COVID-19: Possible mechanisms. Life Sci. 2020 Jul 15;253:117723. doi: 10.1016/j.lfs.2020.117723. Epub 2020 Apr 28. PMID 32360126
- [Result] Xu Z, Shi L, Wang Y, Zhang J, Huang L, Zhang C, Liu S, Zhao P, Liu H, Zhu L, Tai Y, Bai C, Gao T, Song J, Xia P, Dong J, Zhao J, Wang FS. Pathological findings of COVID-19 associated with acute respiratory distress syndrome. Lancet Respir Med. 2020 Apr;8(4):420-422. doi: 10.1016/S2213-2600(20)30076-X. Epub 2020 Feb 18. No abstract available. PMID 32085846
- [Result] Barton LM, Duval EJ, Stroberg E, Ghosh S, Mukhopadhyay S. COVID-19 Autopsies, Oklahoma, USA. Am J Clin Pathol. 2020 May 5;153(6):725-733. doi: 10.1093/ajcp/aqaa062. PMID 32275742
- [Result] Agewall S, Beltrame JF, Reynolds HR, Niessner A, Rosano G, Caforio AL, De Caterina R, Zimarino M, Roffi M, Kjeldsen K, Atar D, Kaski JC, Sechtem U, Tornvall P; WG on Cardiovascular Pharmacotherapy. ESC working group position paper on myocardial infarction with non-obstructive coronary arteries. Eur Heart J. 2017 Jan 14;38(3):143-153. doi: 10.1093/eurheartj/ehw149. No abstract available. PMID 28158518
- [Result] Imazio M, Klingel K, Kindermann I, Brucato A, De Rosa FG, Adler Y, De Ferrari GM. COVID-19 pandemic and troponin: indirect myocardial injury, myocardial inflammation or myocarditis? Heart. 2020 Aug;106(15):1127-1131. doi: 10.1136/heartjnl-2020-317186. Epub 2020 Jun 4. PMID 32499236
- [Result] Wu Z, McGoogan JM. Characteristics of and Important Lessons From the Coronavirus Disease 2019 (COVID-19) Outbreak in China: Summary of a Report of 72 314 Cases From the Chinese Center for Disease Control and Prevention. JAMA. 2020 Apr 7;323(13):1239-1242. doi: 10.1001/jama.2020.2648. No abstract available. PMID 32091533
- [Derived] Filippetti L, Pace N, Louis JS, Mandry D, Goehringer F, Rocher MS, Jay N, Selton-Suty C, Hossu G, Huttin O, Marie PY. Long-Lasting Myocardial and Skeletal Muscle Damage Evidenced by Serial CMR During the First Year in COVID-19 Patients From the First Wave. Front Cardiovasc Med. 2022 Mar 9;9:831580. doi: 10.3389/fcvm.2022.831580. eCollection 2022. PMID 35355964